CLINICAL TRIAL: NCT05524467
Title: RELIEF CENSUS-EU: Cross-sectional Study to Assess Prevalence and Burden of CKD-associated Pruritus in Haemodialysis Patients
Brief Title: Cross-sectional Study to Assess Prevalence and Burden of CKD-associated Pruritus in Haemodialysis Patients
Acronym: ReliefCensus
Status: Completed | Type: Observational
Sponsor: Vifor (International) Inc. (Industry)
Responsible Party: Sponsor
Organization: Vifor Pharma (Industry)
Other Study IDs: CS-DFK-2021-0712
Record Dates: First submitted 2022-08-29; First posted 2022-09-01 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2023-12

CONDITIONS: Chronic Kidney Disease-associated Pruritus
Keywords: CKD; CKD-AP; CKD associated pruritus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Haemodialysis Patients: Only one data collection timepoint per patient is planned. Eligible and consenting patients will be asked to complete several PROs and one questionnaire, and their respective medical charts will be assessed retrospectively

SUMMARY:
Vifor International Inc. is seeking real-world evidence (RWE) to better understand the epidemiology, patient characteristics, and management of CKD-aP in the real-world clinical setting.

DETAILED DESCRIPTION:
This is a non-interventional, cross-sectional, multicentre, and multinational (European) study. The non-interventional study (NIS) design allows the observation of patients in large haemodialysis (HD) centres reflecting routine clinical practice. All decisions on therapeutic or diagnostic procedures, treatments, management of the disease, or resource utilisation will be at the full discretion of the treating physician without interference by the sponsor or study protocol. All treatment decisions will follow the real-life treatment behaviour.

The CENSUS-EU represents a cross-sectional study design of a representative selection of patients undergoing HD at 113 large dialysis centres across 7 countries in Europe. Prot. v.2.0, 9 May 2023

ELIGIBILITY:
Inclusion Criteria:

* Male or female adult patients with CKD (≥18 years) receiving HD for at least 3 months prior to signing informed consent
* Signed informed consent
* Able and willing to fill in questionnaires

Exclusion Criteria:

* Patients performing HD at home or both home and centre

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The CENSUS-EU represents a cross-sectional study design of a representative selection of patients undergoing HD at 113 large dialysis centres across 7 countries in Europe. Prot. v.2.0, 9 May 2023
Sampling Method: Probability Sample
Enrollment: 3100 (Actual)
Dates: Start 2023-02-02 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Prevalence of CKD-aP in HD patients | A 7-month study timeline
  Percentage (%)

SECONDARY OUTCOMES:
The prevalence of CKD-aP by severity | A 7-month study timeline
  none, mild, moderate, and severe

CONTACTS AND LOCATIONS:
Overall Officials: James Burton, Prof., Principal Investigator — University of Leicester Leicester, United Kingdom
Locations (94):
- Germany (17):
  - 1113, Aschaffenburg
  - 1011, Balingen
  - 1007, Braunschweig
  - 1016, Einbeck
  - 1012, Eisenach
  - 1043, Flensburg
  - 1048, Freiburg im Breisgau
  - 1049, Freiburg im Breisgau
  - 1046, Hanover
  - 1001, Herne
  - 1035, Kiel
  - 1111, Leipzig
  - 1013, Mainz
  - 1047, Saalfeld
  - 1053, Sömmerda
  - 1044, Witten
  - 1051, Wuppertal
- Italy (25):
  - 4027, Acquaviva delle Fonti
  - 4015, Bari
  - 4010, Civitavecchia
  - 4001, Florence
  - 4005, Lecce
  - 4016, L’Aquila
  - 4008, Macerata
  - 4023, Mestre
  - 4006, Milan
  - 4018, Milan
  - 4021, Milan
  - 4011, Modena
  - 4009, Monza
  - 4003, Palermo
  - 4017, Parma
  - 4006, Pavia
  - 4028, Pisa
  - 4002, Pistoia
  - 4026, Reggio Calabria
  - 4014, Roma
  - 4024, Rome
  - 4022, Treviso
  - 4030, Trieste
  - 4012, Verona
  - 4025, Viterbo
- Portugal (7):
  - 5014, Cascais
  - 5001, Faro
  - 5013, Gandra
  - 5011, Gondomar
  - 5006, Leiria
  - 5008, Porto
  - 5002, Sacavém
- Spain (25):
  - 3009, Palma de Mallorca, Mallorca
  - 3006, Almería
  - 3005, Barcelona
  - 3011, Barcelona
  - 3012, Barcelona
  - 3026, Barcelona
  - 3002, Benidorm
  - 3008, Cadiz
  - 3001, Gijón
  - 3018, Granada
  - 3025, Jaén
  - 3020, Las Palmas
  - 3021, León
  - 3015, Madrid
  - 3016, Madrid
  - 3022, Madrid
  - 3024, Madrid
  - 3017, Pamplona
  - 3013, Santander
  - 3007, Seville
  - 3023, Seville
  - 3010, Terrassa
  - 3003, Valencia
  - 3004, Valencia
  - 3027, Valencia
- Sweden (8):
  - 6008, Linköping
  - 6007, Malmo
  - 6005, Norrköping
  - 6004, Örebro
  - 6001, Stockholm
  - 6003, Trollhättan
  - 6006, Umeå
  - 6002, Uppsala
- Switzerland (5):
  - 2009, Baden
  - 2001, Bern
  - 2002, Frauenfeld
  - 2004, Lugano
  - 2003, Zurich
- United Kingdom (7):
  - 7002, Bradford
  - 7003, Hull
  - 7001, Leicester
  - 7006, London
  - 7007, London
  - 7005, Nottingham
  - 7004, Sheffield

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be requested 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later.
  Data will be indefinitely available for requesting
Access Criteria: A research proposal must be approved by an independent review panel and the study sponsor and researchers must sign a data sharing agreement.